CLINICAL TRIAL: NCT03219554
Title: Samsung Medical Center
Brief Title: A Phase II Study of Palbociclib for Recurrent or Refractory Advanced Thymic Epithelial Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, MD,PhD,Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-006
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Thymic Cancer
MeSH Terms: conditions — Thymus Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- palbociclib (Experimental): oral palbociclib 125mg daily for 21days followed by a 7-day break. Cycle will be repeated every 28 days.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — oral palbociclib 125mg daily for 21days followed by a 7-day break. Cycle will be repeated every 28 days.

SUMMARY:
This is a phase II single center, open-label, single arm study of palbociclib treatment in patients with recurrent or metastatic advanced TETs after failure of one or more cytotoxic chemotherapy regimens. Patients will receive oral palbociclib 125mg daily for 21days followed by a 7-day break. Cycle will be repeated every 28 days.

DETAILED DESCRIPTION:
Patients will continue to receive Palbociclib until objective disease progression, symptomatic deterioration, unacceptable toxicity, death, or withdrawn of consent, whichever occurs first.

Disease assessments will be performed every 8 weeks (±7 days) from the date of initiation of treatment. Each assessment will be performed as scheduled according to the calendar regardless of any dosing delay to prevent the introduction of bias into the assessment of efficacy. Tumor assessments will be performed until radiographically and/or clinically (ie, for photographed or palpable lesions) documented progressive disease (PD) as per RECIST v.1.1, initiation of new anticancer therapy, or discontinuation of patient from overall study participation (eg, death, patient's request, lost to follow-up), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven thymic epithelial tumor (TET) patients
2. Be ≥18 years of age on day of signing informed consent.
3. Documented progressive disease according to RECIST v1.1 following receipt of at least one cytotoxic chemotherapy regimen administered for inoperable or metastatic disease.
4. Measurable disease as defined per RECIST v 1.1. Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measurable if disease progression at the treated sited after completion of therapy is clearly documented.
5. Availability of a tumor tissue specimen (ie, archived formalin fixed paraffin embedded tissue [block preferred, or 10 unstained slides]), which will be used for retrospective biomarker analysis. If archived tumor tissue is not available, then a de novo biopsy will be required for patient participation.
6. ECOG performance status of 0 to 2

Exclusion Criteria:

1. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (eg, radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
2. Inability to swallow capsules.
3. Prior treatment with any CDK4/6 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival ( PFS) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea